CLINICAL TRIAL: NCT05151289
Title: Diagnostic Value of sFlt-1/PlGF Ratio for the Etiology of Intra Uterine Growth Restriction
Brief Title: Diagnostic Value of sFlt-1/PlGF Ratio for the Etiology of Intra Uterine Growth Restriction - ANGIOPAG
Acronym: ANGIOPAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190472; 2019-A01116-51 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-10-11; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-08

CONDITIONS: Intrauterine Growth Restriction; Fetal Growth Restriction (FGR)
Keywords: sFlt1; PlGF; IUGR; intrauterine growth restriction; fetal growth restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: Patients consulting in one of the participating centers for intra uterine growth restriction.
Masking Description: Regarding the placenta study : for each patient included, the placenta is sent to anatomo-pathology and a referent anatomo-pathologist designated for the study in each center makes an analysis (blind of dosages of sFlt-1/PlGF but not of the clinic)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients consulting in one of the participating centers for intra uterine growth restriction. (Experimental): All included patients
  Interventions: Biological: Blood test at time of inclusion for sFlt-1/PlGF ratio; Biological: Follow-up blood test 2 to 4 weeks after inclusion; Diagnostic Test: Placenta analysis for all included patients, even in case of normal birthweight

INTERVENTIONS:
Biological: Blood test at time of inclusion for sFlt-1/PlGF ratio — As part of the research, a blood sample is taken to measure the sFLT-1 and PlGF ratio at the inclusion visit.
Biological: Follow-up blood test 2 to 4 weeks after inclusion — As part of the research, a blood sample is taken to measure the sFLT-1 and PlGF ratio at the follow-up visit (about 2-4 weeks after inclusion). This second sample is not mandatory for the evaluation of the study's main endpoint.
Diagnostic Test: Placenta analysis for all included patients, even in case of normal birthweight — After delivery, the placenta of each included patient is sent to anatomo-pathology (even in case of normal weight of the baby at birth). An anatomopathologist referent, designated for the study in each center, performs an analysis (aware of the clinic but not of the sFLT-1/PlGF ratio results), according to the benchmark criteria grid. Local analysis will classify the placenta as "vascular IUGR" or "nonvascular IUGR".

SUMMARY:
The main aim of this project is to determine the Placental Growth Factor and Vascular Endothelial Growth Factor ratio's performance (sFlt-1/PlGF) for the etiological diagnosis of vascular Intrauterine growth restriction (IUGR) compared to a non-vascular IUGR.

DETAILED DESCRIPTION:
Intra-uterine growth restriction is one of the most frequent cause of consultation in prenatal diagnosis centers. Suspected Intrauterine growth restriction (IUGR) concerns 5.4% of pregnancies. Prognosis and management of IUGR depends on its etiology. It has been estimated that 80 to 90% of IUGR have a vascular cause, 5-15% an infectious cause and 2 to 5% chromosomal or genetic cause. More recently, a meta-analysis has shown that among 874 IUGR fetuses for whom amniocentesis was performed, anomaly of caryotype or comparative genomic hybridization array was reported for 6%. In case of vascular IUGR, amniocentesis is not indicated and close surveillance of mother and fetus is organized.

The diagnosis of vascular IUGR is most often confirmed after birth with placental histology. Before birth, the diagnosis of vascular IUGR is presumptive, and based on gestational age at diagnosis, quantity of amniotic fluid, end dopplers of umbilical artery and uterine arteries. The argument considered as most specific of vascular IUGR is the doppler of uterine arteries, however it has been shown that sensitivity of this test is weak : abnormal uterine arteries is reported in only 40% of fetuses with vasculat IUGR according to placenta pathology.

Biochemical markers Placental Growth Factor and Vascular Endothelial Growth Factor (sFlt1 and PlGF) have shown their prognostic value on the occurrence of preeclampsia. They are both associated to the delay until occurrence of preeclampsia and to the delay before extraction in case of IUGR. As diagnostic tool in IUGR, only two studies have investigated their value : the PlGF/sFlt-1 ratio identified 7 patients among 10 with abnormal placental pathology, and low PlGF value is associated with abnormal placental pathology among 122 cases of IUGR, however this study did not specify sensitivity and specificity values. A reliable and reproductible marker that could orient practitioners towards the need to propose amniocentesis at diagnosis of IUGR is therefore important to develop.

The main objective of ANGIOPAG is to determine the sFlt-1/PlGF ratio's performance for the etiological diagnosis of vascular IUGR compared to a non-vascular IUGR.

To reach this goal, ANGIOPAG is a diagnostic, multicenter, non-randomized study. It will be performed on 152 pregnant women over 18 with a term between 22and 34 +6 Weeks of Gestation (WG), consulting in participating centers for IUGR. For the research, a blood test will be carried, at the inclusion and 2 to 4 weeks after, to determine sFLT-1 and PlGF. All included patients'placenta will be analyzed, even in case of a child normal birth weight.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Singleton pregnancy
* Date of conception evaluated by ultrasound < 14 WG
* Consulting in one of the 3 participating centers for IUGR
* Estimated fetal weight < 5th centile (according to Hadlock 3 et CFEF)
* Between 22+0 WG et 34+6 WG

Exclusion Criteria:

* Major birth defect diagnosed at time of inclusion
* Abnormality of caryotype known at time of inclusion
* Confirmed preeclampsia at time of inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-01-29 (Estimated); Study Completion 2022-01-29 (Estimated)

PRIMARY OUTCOMES:
To compare the PlGF / sFlt-1 ratio and placental lesions to confirm the diagnosis of vascular intrauterine growth retardation | 34+6 Weeks of Gestation
  The etiological diagnosis will be confirmed as vascular if characteristic lesions are identified on placental analysis. Lesions of maternal vascular malperfusion have been described and are those used in scientific literature. These characteristics are placental infarcts, decidual arteriopathy, and villous hypoplasia.

SECONDARY OUTCOMES:
Delay between inclusion and birth | 21 weeks after inclusion
  Delay between inclusion and birth
Occurrence of preeclampsia | 21 weeks after inclusion
  Occurrence of preeclampsia
Gestational age at birth | maximum 21 weeks after inclusion
  Gestational age at birth
Birth weight | maximum 21 weeks after inclusion
  Birth weight
Newborn evaluation (presence of birth defects) | maximum 21 weeks after inclusion
  Newborn evaluation (presence of birth defects)
Rate of transfers to intensive care unit | maximum 21 weeks after inclusion
  Rate of transfers to intensive care unit
Rate of death of babies | maximum 21 weeks after inclusion
  Rate of death of babies

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Sibiude, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Colombes, France